CLINICAL TRIAL: NCT02449941
Title: Distribution of Helicobacter Pylori According to the Use of Proton Pump Inhibitor
Brief Title: Helicobacter Pylori and Proton Pump Inhibitor
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Yong Ahn, Professor, Asan Medical Center
Other Study IDs: 2014-0341
Record Dates: First submitted 2015-05-14; First posted 2015-05-21 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Helicobacter Infections
Keywords: Stomach Neoplasms; proton pump inhibitor; endoscopic submucosal dissection; Helicobacter pylori; Gastritis, Atrophic
MeSH Terms: conditions — Helicobacter Infections; Stomach Neoplasms; Gastritis, Atrophic | interventions — Proton Pump Inhibitors; Pantoprazole; Lansoprazole; Dexlansoprazole; Rabeprazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — endoscopic biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Helicobacter pylori(HP) positive: Participants who are diagnosed with Helicobacter Pylori infection through ESD(endoscopic submucosal dissection) will be treated with PPI (proton pump inhibitor).
  Interventions: Drug: PPI (proton pump inhibitor)

INTERVENTIONS:
Drug: PPI (proton pump inhibitor) — 1. Pre ESD (endoscopic submucosal dissection)
     * Assessment atrophy and metaplasia in stomach, Check Helicobacter pylori
     * Use of PPI for 2 months
  2. Post ESD 1 (After 2 months)
     * Assess the distribution of helicobacter pylori after using PPI.
     * Stop of PPI
  3. Post ESD 2 (After 4 months)
     * Assess the distribution of helicobacter pylori after stop of PPI.
  Other Names: pantoprazole, lansoprazole, dexlansoprazole, rabeprazole

SUMMARY:
The purpose of this study is to know the distribution of HP in stomach before use of PPI, during use of PPI, and after stop of PPI.

DETAILED DESCRIPTION:
Endoscopy and biopsy will be performed to investigate the distrubition of HP before, during, and after using PPI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are indicated to endoscopic resection due to gastric neoplasm
2. Aged between 19 to 65 years
3. Informed consent

Exclusion Criteria:

1. Previous history of HP eradication
2. Previous history of PPI use within 6 months
3. No HP infection

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample size will be determined based on the analysis the distribution rate of HP at first 30 patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Analysis the change of Helicobacter pylori distribution according to the use of proton pump inhibitor | Change in the distribution of Helicobacter Pylori(HP) at 4 months.

SECONDARY OUTCOMES:
Analysis the change of HP distribution according to the use of PPI in atrophic change of stomach | Change in the distribution of Helicobacter Pylori(HP) at 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Yong Ahn, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong EJ, Kim DH, Ahn JY, Na HK, Jung KW, Lee JH, Choi KD, Song HJ, Lee GH, Jung HY, Park Y, Kim MJ. Effects of Proton Pump Inhibitor on the Distribution of Helicobacter pylori and Associated Gastritis in Patients with Gastric Atrophy. Digestion. 2020;101(3):279-286. doi: 10.1159/000499424. Epub 2019 May 8. PMID 31067538